CLINICAL TRIAL: NCT04046939
Title: A Randomized, Double-Blind, Placebo-Controlled Dose-Ranging Biomarker Study of the Effects of Dexpramipexole on Eosinophils in Subjects With Eosinophilic Asthma
Brief Title: Dexpramipexole Dose-Ranging Biomarker Study in Subjects With Eosinophilic Asthma
Acronym: EXHALE-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Knopp Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KNS-760704-AS201
Record Dates: First submitted 2019-07-30; First posted 2019-08-06 (Actual); Results first posted 2021-12-22 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Eosinophilic Asthma; Asthma
Keywords: Eosinophilic Asthma; Asthma; dexpramipexole
MeSH Terms: conditions — Pulmonary Eosinophilia; Asthma | interventions — Dexpramipexole

STUDY DESIGN:
Intervention Model Description: Four-arm parallel assignment
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- placebo BID (Placebo Comparator): Following a 2-4 week placebo run-in, randomized subjects received 1 tablet placebo twice daily for 12 weeks.
  Interventions: Drug: Placebo
- 37.5 mg BID dexpramipexole (Active Comparator): Following a 2-4 week placebo run-in, randomized subjects received 1 tablet of 37.5 mg dexpramipexole twice daily for 12 weeks.
  Interventions: Drug: Dexpramipexole
- 75 mg BID dexpramipexole (Active Comparator): Following a 2-4 week placebo run-in, randomized subjects received 1 tablet of 75 mg dexpramipexole twice daily for 12 weeks.
  Interventions: Drug: Dexpramipexole
- 150 mg BID dexpramipexole (Active Comparator): Following a 2-4 week placebo run-in, randomized subjects received 1 tablet of 150 mg dexpramipexole twice daily for 12 weeks.
  Interventions: Drug: Dexpramipexole

INTERVENTIONS:
Drug: Dexpramipexole — dexpramipexole twice daily oral dosing for up to 12 weeks
  Other Names: KNS-760704; BIIB050
  Arms: 150 mg BID dexpramipexole; 37.5 mg BID dexpramipexole; 75 mg BID dexpramipexole
Drug: Placebo — placebo twice daily oral dosing for up to 12 weeks
  Other Names: PBO
  Arms: placebo BID

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group, dose-ranging, multi-center study to evaluate the clinical effects of oral administration of dexpramipexole for 12 weeks on peripheral blood eosinophil count in subjects with eosinophilic asthma.

DETAILED DESCRIPTION:
One hundred subjects will receive study drug or matching placebo over 12 weeks of consecutive dosing. Following a short Run-in Period, eligible subjects will enter the Primary Assessment Period and receive twice-daily dosing of study drug or placebo for 12 weeks. Following 12 weeks of treatment, subjects will enter a 12-week Eosinophil Recovery Period. The primary endpoint for the study is the change in blood absolute eosinophil count from Baseline to Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 and <75 years of age at the time of consent
* Physician diagnosis of asthma for ≥12 months (relative to Baseline) based on Global Initiative for Asthma (GINA) 2018 Guidelines
* Asthma requiring treatment with, at a minimum, low dose inhaled corticosteroids in combination with a long-acting β2 agonist, on a stable dose for at least 1 month before Screening
* Bronchodilator reversibility, as evidenced by ≥12% and ≥200 mL improvement in FEV1 15 to 25 minutes following inhalation of albuterol at Screening
* Pre-bronchodilator FEV1 ≥40% and <80% of predicted at Screening and Baseline
* AEC ≥0.30 x10^9/L at the Screening visit
* ACQ-7 ≥1.5 at Screening
* Negative pregnancy test at Baseline
* Adherence ≥85% with twice-daily placebo taken during the Run-in Period

Exclusion Criteria:

* Treatment for an asthma exacerbation within 8 weeks prior to Baseline visit
* Treatment with systemic corticosteroids in the 8 weeks prior to Screening
* Treatment with monoclonal antibody therapy, within 5-half-lives prior to Baseline
* Treatment with selected drugs known to have a substantial risk of neutropenia
* Absolute neutrophil count <2.0x10^9/L at Screening, or any documented history of absolute neutrophil count <2.0x10^9/L.
* Renal dysfunction, defined as an estimated glomerular filtration rate (eGFR) <60 mL/min/1.73m^2 at Screening
* Clinically significant abnormal laboratory or ECG values
* Other medically significant illness
* Use of any smoke or inhaled nicotine delivery device within 1 year prior to Screening
* Pregnant women or women breastfeeding
* Currently taking pramipexole or other dopamine agonists

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 534 (Actual)
Dates: Start 2019-08-15 (Actual); Primary Completion 2020-12-03 (Actual); Study Completion 2021-03-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (33):
  - Research Site, Los Angeles, California
  - Research Site, Mission Viejo, California
  - Research Site, Westminster, California
  - Research Site, Denver, Colorado
  - Research Site, Daytona Beach, Florida
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Tampa, Florida
  - Research Site, Lawrenceville, Georgia
  - Research Site, Winder, Georgia
  - Research Site, Boise, Idaho
  - Research Site, Farmington Hills, Michigan
  - Research site, Plymouth, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, Las Vegas, Nevada
  - Research Site, New Brunswick, New Jersey
  - Research Site, Corning, New York
  - Research Site, New Hyde Park, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Dublin, Ohio
  - Research Site, Edmond, Oklahoma
  - Research Site, Medford, Oregon
  - Research Site, Portland, Oregon
  - Research Site, Pittsburgh, Pennsylvania
  - Research Site, Anderson, South Carolina
  - Research Site, North Charleston, South Carolina
  - Research Site, Allen, Texas
  - Research Site, Boerne, Texas
  - Research Site, Dallas, Texas
  - Research Site, El Paso, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 534 participants enrolled, 144 subjects received placebo treatment during the Run-in Period. Of those, 103 completed the Run-in Period, were eligible for randomization, and entered the Primary Assessment Period.
Period: Screening Period
Arm/Group | Placebo BID | 37.5 mg BID Dexpramipexole | 75 mg BID Dexpramipexole | 150 mg BID Dexpramipexole
Started | 534 | 0 | 0 | 0
Received Placebo During Run-In Period | 144 | 0 | 0 | 0
Completed | 103 | 0 | 0 | 0
Not Completed | 431 | 0 | 0 | 0
Period: Primary Assessment Period
Arm/Group | Placebo BID | 37.5 mg BID Dexpramipexole | 75 mg BID Dexpramipexole | 150 mg BID Dexpramipexole
Started | 27 | 22 | 26 | 28
Completed | 25 | 22 | 24 | 28
Not Completed | 2 | 0 | 2 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Period: Eosinophil Recovery Period
Arm/Group | Placebo BID | 37.5 mg BID Dexpramipexole | 75 mg BID Dexpramipexole | 150 mg BID Dexpramipexole
Started | 25 | 22 | 24 | 28
Completed | 24 | 22 | 24 | 27
Not Completed | 1 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population: all subjects who were randomized and received at least 1 dose of study drug (placebo, dexpramipexole) during the Primary Assessment Period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo BID | 37.5 mg BID Dexpramipexole | 75 mg BID Dexpramipexole | 150 mg BID Dexpramipexole | Total
Number analyzed (Participants) | 27 | 22 | 26 | 28 | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (12.89) | 46.6 (13.41) | 44.5 (15.46) | 44.6 (12.53) | 45.3 (13.42)
Age, Customized [Count of Participants; unit: Participants]
  <50 years | 15 | 14 | 15 | 18 | 62
  50 to 65 years | 10 | 6 | 8 | 9 | 33
  >65 years | 2 | 2 | 3 | 1 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 11 | 14 | 12 | 54
  Male | 10 | 11 | 12 | 16 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 3 | 3 | 11
  Not Hispanic or Latino | 25 | 19 | 23 | 25 | 92
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 1 | 2 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 4 | 4 | 6 | 6 | 20
  White | 21 | 17 | 16 | 22 | 76
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Body mass index (kg/m^2) = body weight (kg) / height (m^2)
  kg/m^2 | 34.31 (12.749) | 31.73 (7.379) | 33.44 (10.690) | 32.13 (7.040) | 32.95 (9.738)

OUTCOME MEASURES:

1. Primary Outcome: Change in Blood Absolute Eosinophil Count From Baseline to Week 12
Description: The primary endpoint of this study was the change in AEC from Baseline to Week 12 on a ratio scale. The analysis used a mixed effects model repeated-measures (MMRM) with terms for log10 transformed baseline, GINA treatment step, treatment, visit, treatment by visit interaction, and log10 transformed baseline by visit interaction as fixed effects, and subject as a random effect. An unstructured covariance matrix was used. The response variable was the log10 transformed post-baseline value minus the log10 transformed baseline value. The estimates of Geometric LS Means and their ratios were obtained by back transforming the corresponding estimates of LS means and their differences to the original scale.
Time Frame: Baseline, 12 Weeks
Population: The efficacy population will be a modified intent-to-treat sample and consist of all subjects in the safety population (all subjects who were randomized and received at least one dose of randomized study drug) and who have at least one post-randomization AEC evaluation.
Measure: Geometric Least Squares Mean (Standard Error); unit: ratio to baseline
Arm/Group | Placebo BID | 37.5 mg BID Dexpramipexole | 75 mg BID Dexpramipexole | 150 mg BID Dexpramipexole
Number analyzed (Participants) | 25 | 22 | 24 | 28
ratio to baseline | 0.8980 (1.26) | 0.4031 (1.28) | 0.3056 (1.27) | 0.2051 (1.25)
Statistical Analysis 1: Comparison: Placebo BID vs 150 mg BID Dexpramipexole; The 150 mg BID dexpramipexole group was compared to placebo using a mixed effects model repeated-measures (MMRM); Test type: Superiority; p < .0001, Mixed Models Analysis — A closed hierarchical procedure testing dexpramipexole against placebo at Week 12 was used. (1) 150 mg BID for AEC (2) 75 mg BID for AEC (3) pooled 75 mg and 150 mg BID group for pre-bronchodilator FEV1; and (4) 37.5 mg BID for AEC; Ratio to PBO of the ratios to baseline = 0.2283, 95% CI 2-sided [0.121 to 0.431] — 0.2283 represents the ratio of the 150 mg BID week 12 ratio to baseline (0.2051), compared to the PBO week 12 ratio to baseline (0.8980). This ratio of 0.2283 is equivalent to a -77.17% change compared to placebo at week 12
Statistical Analysis 2: Comparison: Placebo BID vs 75 mg BID Dexpramipexole; The 75 mg BID dexpramipexole group was compared to placebo using a mixed effects model repeated-measures (MMRM); Test type: Superiority; p = 0.0014, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Ratio to PBO of the ratios to baseline = 0.3403, 95% CI 2-sided [0.177 to 0.653] — 0.3403 represents the ratio of the 75 mg BID week 12 ratio to baseline (0.3056), compared to the PBO week 12 ratio to baseline (0.8980). This ratio of 0.3403 is equivalent to a -65.97% change compared to placebo at week 12
Statistical Analysis 3: Comparison: Placebo BID vs 37.5 mg BID Dexpramipexole; The 37.5 mg BID dexpramipexole group was compared to placebo using a mixed effects model repeated-measures (MMRM); Test type: Superiority; p = 0.0190, Mixed Models Analysis — A closed hierarchical statistical testing was used. The previous endpoint in the hierarchy was not statistically significant. Therefore, this endpoint was not formally tested and is not considered statistically significant, despite a p-value <0.05; Ratio to PBO of the ratios to baseline = 0.4489, 95% CI 2-sided [0.231 to 0.874] — 0.4489 represents the ratio of the 37.5 mg BID week 12 ratio to baseline (0.4031) compared to the PBO week 12 ratio to baseline (0.8980). This ratio of 0.4489 is equivalent to a -55.11% change compared to placebo at week 12

2. Secondary Outcome: Change in Pre-bronchodilator FEV1 (Liters) From Baseline to Week 12
Description: FEV1 is defined as the amount of air that can be forcibly exhaled from the lungs in the first second of a forced exhalation.
Time Frame: Baseline, 12 Weeks
Population: The efficacy population will be a modified intent-to-treat sample and consist of all subjects in the safety population (all subjects who were randomized and received at least one dose of randomized study drug) and who have at least one post-randomization FEV1 evaluation. Spirometry restrictions were put in place during the COVID-19 pandemic. Subjects who did not complete the Week 8 and Week 12 post dose assessments due to these restrictions were excluded from this analysis.
Measure: Least Squares Mean (Standard Error); unit: liters
Groups:
- Combined 150 mg BID and 75 mg BID Arms: Following a 2-4 week placebo run-in, randomized subjects in this combined treatment group received 1 tablet of either 150 mg dexpramipexole twice daily for 12 weeks or 75 mg dexpramipexole trice daily for 12 weeks.
  Dexpramipexole: dexpramipexole twice daily oral dosing for up to 12 weeks
Arm/Group | Placebo BID | 37.5 mg BID Dexpramipexole | 75 mg BID Dexpramipexole | 150 mg BID Dexpramipexole | Combined 150 mg BID and 75 mg BID Arms
Number analyzed (Participants) | 17 | 18 | 21 | 24 | 45
liters | 0.0700 (0.08329) | 0.208 (0.08387) | 0.0557 (0.07848) | 0.247 (0.07769) | 0.151 (0.05746)
Statistical Analysis 1: Comparison: Placebo BID vs Combined 150 mg BID and 75 mg BID Arms; The combined 75 mg and 150 mg BID dexpramipexole group was compared to placebo using a mixed effects model repeated-measures (MMRM); Test type: Superiority; p = 0.4154, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.0814, 95% CI 2-sided [-0.116 to 0.279] — Estimate is the difference of the pooled 75 mg and 150 mg BID group from placebo in change in pre-bronchodilator FEV1 in liters from Baseline to Week 12 (end of primary treatment period). A positive value indicates improvement in lung function
Statistical Analysis 2: Comparison: Placebo BID vs 150 mg BID Dexpramipexole; The 150 mg BID dexpramipexole group was compared to placebo using a mixed effects model repeated-measures (MMRM); Test type: Superiority; p = 0.1174, Mixed Models Analysis — For secondary endpoints which were not key secondary endpoints, no adjustment for multiple testing was used and p <0.05 was used for statistical significance; Mean Difference (Final Values) = 0.177, 95% CI 2-sided [-0.0456 to 0.400] — Estimate is the difference of the 150 mg BID group from the placebo group in the change in pre-bronchodilator FEV1 in liters from Baseline to Week 12 (end of primary treatment period). A positive value indicates improvement in lung function
Statistical Analysis 3: Comparison: Placebo BID vs 75 mg BID Dexpramipexole; The 75 mg BID dexpramipexole group was compared to placebo using a mixed effects model repeated-measures (MMRM); Test type: Superiority; p = 0.8998, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; Mean Difference (Final Values) = -0.0143, 95% CI 2-sided [-0.240 to 0.211] — Estimate is the difference of the 75 mg BID group from the placebo group in the change in pre-bronchodilator FEV1 in liters from Baseline to Week 12 (end of primary treatment period). A positive value indicates improvement in lung function
Statistical Analysis 4: Comparison: Placebo BID vs 37.5 mg BID Dexpramipexole; The 37.5 mg BID dexpramipexole group was compared to placebo using a mixed effects model repeated-measures (MMRM); Test type: Superiority; p = 0.2425, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; Mean Difference (Final Values) = 0.138, 95% CI 2-sided [-0.0950 to 0.370] — Estimate is the difference of the 37.5 mg BID group from the placebo group in the change in pre-bronchodilator FEV1 in liters from Baseline to Week 12 (end of primary treatment period). A positive value indicates improvement in lung function

3. Secondary Outcome: Change in Asthma Control Questionnaire (ACQ-6) Score From Baseline to Week 12
Description: ACQ-6 is simple questionnaire to measure the adequacy of asthma control and change in asthma control which occurs either spontaneously or as a result of treatment. The 6-point self-administered scale has items measuring asthma symptoms and rescue inhaler use. The ACQ score is the mean of the questions and therefore between 0 (totally controlled) and 6 (severely uncontrolled). The original protocol planned to analyze the ACQ-7 score. As a result of FEV1 testing restrictions imposed on the study during the COVID-19 pandemic, the analysis was prospectively modified to the ACQ-6 score prior to database lock. The ACQ-6 is a validated questionnaire and is identical to the ACQ-7, with the exception of FEV1 data that is also utilized in the ACQ-7 questionnaire total score calculation.
Time Frame: Baseline, 12 Weeks
Population: The efficacy population was a modified intent-to-treat sample and consist of all subjects in the safety population (all subjects who were randomized and received at least one dose of randomized study drug) and who have at least one post-randomization evaluation.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo BID | 37.5 mg BID Dexpramipexole | 75 mg BID Dexpramipexole | 150 mg BID Dexpramipexole
Number analyzed (Participants) | 25 | 22 | 24 | 28
scores on a scale | -0.391 (0.1866) | -0.419 (0.1974) | -0.437 (0.1924) | -0.655 (0.1803)
Statistical Analysis 1: Comparison: Placebo BID vs 150 mg BID Dexpramipexole; The 150 mg BID dexpramipexole group was compared to placebo using a mixed effects model repeated-measures (MMRM); Test type: Superiority; p = 0.3059, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; Mean Difference (Final Values) = -0.264, 95% CI 2-sided [-0.772 to 0.245] — Estimate is the difference of the 150 mg BID dexpramipexole group compared to the placebo group in change in ACQ-6 score from Baseline to Week 12 (end of primary treatment period). A negative value indicates improvement of asthma symptoms
Statistical Analysis 2: Comparison: Placebo BID vs 75 mg BID Dexpramipexole; The 75 mg BID dexpramipexole group was compared to placebo using a mixed effects model repeated-measures (MMRM); Test type: Superiority; p = 0.8642, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; Mean Difference (Final Values) = -0.0457, 95% CI 2-sided [-0.575 to 0.484] — Estimate is the difference of the 75 mg BID dexpramipexole group compared to the placebo group in change in ACQ-6 score from Baseline to Week 12 (end of primary treatment period). A negative value indicates improvement of asthma symptoms
Statistical Analysis 3: Comparison: Placebo BID vs 37.5 mg BID Dexpramipexole; The 37.5 mg BID dexpramipexole group was compared to placebo using a mixed effects model repeated-measures (MMRM); Test type: Superiority; p = 0.9182, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 2]; Mean Difference (Final Values) = -0.0276, 95% CI 2-sided [-0.560 to 0.505] — Estimate is the difference of the 37.5 mg BID dexpramipexole group compared to the placebo group in change in ACQ-6 score from Baseline to Week 12 (end of primary treatment period). A negative value indicates improvement of asthma symptoms

4. Secondary Outcome: Change in Post-bronchodilator FEV1 From Baseline to Week 12
Description: Post-bronchodilator FEV1 is defined as the amount of air that can be forcibly exhaled from the lungs in the first second of a forced exhalation, after treatment with inhaled albuterol.
Time Frame: Baseline, 12 Weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo BID | 37.5 mg BID Dexpramipexole | 75 mg BID Dexpramipexole | 150 mg BID Dexpramipexole
Number analyzed (Participants) | 20 | 18 | 22 | 23
liters | -0.00546 (0.07208) | 0.0932 (0.07455) | -0.000717 (0.06977) | 0.176 (0.07182)
Statistical Analysis 1: Comparison: Placebo BID vs 150 mg BID Dexpramipexole; An ANCOVA analysis was performed comparing the 150 mg BID dexpramipexole group to placebo; Test type: Superiority; p = 0.0716, ANCOVA — [p-value comment as in outcome 2, analysis 2]; Mean Difference (Final Values) = 0.181, 95% CI 2-sided [-0.0163 to 0.378] — Estimate the difference of the 150 mg BID Dexpramipexole group from placebo in change in post-bronchodilator FEV1 from Baseline to Week 12 (end of primary treatment period) in liters. A positive value indicates improvement in lung function
Statistical Analysis 2: Comparison: Placebo BID vs 75 mg BID Dexpramipexole; An ANCOVA analysis was performed comparing the 75 mg BID dexpramipexole group to placebo; Test type: Superiority; p = 0.9619, ANCOVA — [p-value comment as in outcome 2, analysis 2]; Mean Difference (Final Values) = 0.00474, 95% CI 2-sided [-0.192 to 0.202] — Estimate the difference of the 75 mg BID Dexpramipexole group from placebo in change in post-bronchodilator FEV1 from Baseline to Week 12 (end of primary treatment period) in liters. A positive value indicates improvement in lung function
Statistical Analysis 3: Comparison: Placebo BID vs 37.5 mg BID Dexpramipexole; An ANCOVA analysis was performed comparing the 37.5 mg BID dexpramipexole group to placebo; Test type: Superiority; p = 0.3368, ANCOVA — [p-value comment as in outcome 2, analysis 2]; Median Difference (Final Values) = 0.0987, 95% CI 2-sided [-0.105 to 0.302] — Estimate the difference of the 37.5 mg BID Dexpramipexole group from placebo in change in post-bronchodilator FEV1 from Baseline to Week 12 (end of primary treatment period) in liters. A positive value indicates improvement in lung function

5. Secondary Outcome: Change in Quality of Life, as Measured by the Asthma Quality of Life Questionnaire (AQLQ) From Baseline to Week 12
Description: The AQLQ is a 32-item asthma specific questionnaire designed to measure functional impairments that are most important to patients with asthma. The 32 questions in the AQLQ are divided into four domains; activity limitations, symptoms, emotional function, and environmental stimuli. Individual questions are equally weighted. The overall AQLQ score is the mean of the responses to each of the 32 questions and ranges from 1 to 7. A score 7.0 indicates that the patient has no impairments due to asthma and score 1.0 indicates severe impairment.
Time Frame: Baseline, 12 Weeks
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo BID | 37.5 mg BID Dexpramipexole | 75 mg BID Dexpramipexole | 150 mg BID Dexpramipexole
Number analyzed (Participants) | 26 | 22 | 25 | 28
scores on a scale | 0.376 (0.1999) | 0.531 (0.2112) | 0.312 (0.2055) | 0.584 (0.1979)
Statistical Analysis 1: Comparison: Placebo BID vs 150 mg BID Dexpramipexole; An ANCOVA analysis was performed comparing the 150 mg BID dexpramipexole group to placebo; Test type: Superiority; p = 0.4512, ANCOVA — [p-value comment as in outcome 2, analysis 2]; Mean Difference (Final Values) = 0.208, 95% CI 2-sided [-0.338 to 0.755] — Estimate the difference in the 150 mg BID dexpramipexole group from the placebo group in the change in AQLQ score from Baseline to Week 12 (end of primary treatment period). A positive value indicates improvement of asthma symptoms
Statistical Analysis 2: Comparison: Placebo BID vs 75 mg BID Dexpramipexole; An ANCOVA analysis was performed comparing the 75 mg BID dexpramipexole group to placebo; Test type: Superiority; p = 0.8214, ANCOVA — [p-value comment as in outcome 2, analysis 2]; Mean Difference (Final Values) = -0.0642, 95% CI 2-sided [-0.627 to 0.499] — Estimate the difference in the 75 mg BID dexpramipexole group from the placebo group in the change in AQLQ score from Baseline to Week 12 (end of primary treatment period). A positive value indicates improvement of asthma symptoms
Statistical Analysis 3: Comparison: Placebo BID vs 37.5 mg BID Dexpramipexole; An ANCOVA analysis was performed comparing the 37.5 mg BID dexpramipexole group to placebo; Test type: Superiority; p = 0.5894, ANCOVA — [p-value comment as in outcome 2, analysis 2]; Mean Difference (Final Values) = 0.154, 95% CI 2-sided [-0.411 to 0.720] — Estimate the difference in the 37.5 mg BID dexpramipexole group from the placebo group in the change in AQLQ score from Baseline to Week 12 (end of primary treatment period). A positive value indicates improvement of asthma symptoms

6. Secondary Outcome: Number of Participants With Potentially Clinically Significant Hematology Results by Treatment Group Post Randomization Through Week 12
Description: Number of Participants with Potentially Clinically Significant Hematology Results by Treatment Group. Percentages based on number of patients with at least one non-missing post-baseline value in each treatment group. Patients are only counted once per criterion per laboratory test.
Time Frame: Immediately post-baseline up to Week 12
Population: The safety population includes all subjects who were randomized and received at least one dose of study drug during the primary treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID | 37.5 mg BID Dexpramipexole | 75 mg BID Dexpramipexole | 150 mg BID Dexpramipexole
Number analyzed (Participants) | 27 | 22 | 26 | 28
Participants
  Eosinophils >1.6 x 10^9/L | 0 | 0 | 0 | 0
  Basophils >1.6 x 10^9/L | 0 | 0 | 0 | 0
  Erythrocytes ≤3.5 x 10^12/L | 0 | 1 | 0 | 2
  Erythrocytes ≥6.4 x 10^12/L | 0 | 0 | 0 | 0
  Hematocrit ≤32% - Females: number analyzed (Participants) | 17 | 11 | 14 | 12
  Hematocrit ≤32% - Females | 0 | 2 | 0 | 1
  Hematocrit ≥54% - Females: number analyzed (Participants) | 17 | 11 | 14 | 12
  Hematocrit ≥54% - Females | 0 | 0 | 0 | 0
  Hematocrit ≤37% - Males: number analyzed (Participants) | 10 | 11 | 12 | 16
  Hematocrit ≤37% - Males | 2 | 0 | 1 | 1
  Hematocrit ≥60% - Males: number analyzed (Participants) | 10 | 11 | 12 | 16
  Hematocrit ≥60% - Males | 0 | 0 | 0 | 0
  Hemoglobin ≤9.5 g/dL - Females: number analyzed (Participants) | 17 | 11 | 14 | 12
  Hemoglobin ≤9.5 g/dL - Females | 0 | 1 | 0 | 0
  Hemoglobin ≥17.5 g/dL - Females: number analyzed (Participants) | 17 | 11 | 14 | 12
  Hemoglobin ≥17.5 g/dL - Females | 0 | 0 | 0 | 0
  Hemoglobin ≤11.5 g/dL - Males: number analyzed (Participants) | 10 | 11 | 12 | 16
  Hemoglobin ≤11.5 g/dL - Males | 2 | 0 | 0 | 1
  Hemoglobin ≥19.0 g/dL - Males: number analyzed (Participants) | 10 | 11 | 12 | 16
  Hemoglobin ≥19.0 g/dL - Males | 0 | 0 | 0 | 0
  Leukocytes <3.0 x 10^9/L | 0 | 0 | 0 | 1
  Leukocytes ≥16 x 10^9/L | 0 | 1 | 0 | 1
  Lymphocytes <0.8 x 10^9/L | 0 | 0 | 0 | 1
  Lymphocytes >12 x 10^9/L | 0 | 0 | 0 | 0
  Monocytes >2.5 x 10^9/L | 0 | 0 | 0 | 0
  Neutrophils <1.5 x 10^9/L | 1 | 1 | 1 | 1
  Neutrophils ≥13.5 x 10^9/L | 0 | 0 | 0 | 0
  Platelets ≤75 x 10^9/L | 0 | 0 | 0 | 0
  Platelets ≥700 x 10^9/L | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Potentially Clinically Significant Blood Chemistry Results by Treatment Group Post Randomization Through Week 12
Description: Number of Participants with Potentially Clinically Significant Blood Chemistry Results by Treatment Group. Percentages based on number of patients with at least one non-missing post-baseline value in each treatment group. Patients are only counted once per criterion per laboratory test.
Time Frame: Immediately post-baseline up to Week 12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID | 37.5 mg BID Dexpramipexole | 75 mg BID Dexpramipexole | 150 mg BID Dexpramipexole
Number analyzed (Participants) | 27 | 22 | 26 | 28
Participants
  ALT ≥ 3 x ULN | 0 | 0 | 1 | 0
  Albumin ≤ 2.5 g/dL | 0 | 0 | 0 | 0
  Alkaline Phosphatase ≥ 1.5 x ULN | 0 | 0 | 1 | 1
  AST ≥ 3 x ULN | 0 | 0 | 0 | 0
  Bicarbonate ≤ 16 mEq/L | 0 | 0 | 1 | 0
  Bicarbonate ≥ 35 mEq/L | 0 | 0 | 0 | 0
  Bilirubin > 2 X ULN and (ALT or AST ≥ 3 X ULN) | 0 | 0 | 0 | 0
  Bilirubin ≥ 1.5 x ULN | 0 | 0 | 0 | 0
  Calcium ≤ 8 mg/dL | 0 | 2 | 0 | 3
  Calcium ≥ 12 mg/dL | 0 | 0 | 0 | 0
  Chloride ≤ 90 mEq/L | 0 | 0 | 0 | 0
  Chloride ≥ 118 mEq/L | 0 | 0 | 0 | 0
  Creatinine ≥ 2 mg/dL - Females: number analyzed (Participants) | 17 | 11 | 14 | 12
  Creatinine ≥ 2 mg/dL - Females | 0 | 0 | 0 | 0
  Creatinine ≥ 2 mg/dL - Males: number analyzed (Participants) | 10 | 11 | 12 | 16
  Creatinine ≥ 2 mg/dL - Males | 0 | 0 | 0 | 0
  Glucose ≤ 39.6 mg/dL | 0 | 0 | 0 | 0
  Glucose ≥ 175 mg/dL | 2 | 2 | 1 | 1
  Magnesium ≤ 1.2 mg/dL | 0 | 1 | 0 | 1
  Magnesium ≥ 2.9 mg/dL | 0 | 0 | 0 | 0
  Phosphate ≤ 1.86 mg/dL | 0 | 0 | 0 | 0
  Phosphate ≥ 5.27 mg/dL | 0 | 0 | 0 | 0
  Potassium ≤ 3 mEq/L | 0 | 0 | 0 | 0
  Potassium ≥ 6 mEq/L | 0 | 0 | 0 | 0
  Protein [Serum] ≤ 4.5 g/dL | 0 | 0 | 0 | 0
  Protein [Serum] ≥ 10 g/dL | 0 | 0 | 0 | 0
  Sodium ≤ 126 mEq/L | 0 | 0 | 0 | 0
  Sodium ≥ 156 mEq/L | 0 | 0 | 0 | 0
  Urate ≥ 8.5 mg/dL - Females: number analyzed (Participants) | 17 | 11 | 14 | 12
  Urate ≥ 8.5 mg/dL - Females | 0 | 0 | 0 | 1
  Urate ≥ 10.5 mg/dL - Males: number analyzed (Participants) | 10 | 11 | 12 | 16
  Urate ≥ 10.5 mg/dL - Males | 0 | 0 | 0 | 0
  Urea Nitrogen ≥ 30 mg/dL | 0 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Potentially Clinically Significant Urinalysis Results by Treatment Group Post Randomization Through Week 12
Description: Number of Participants with Potentially Clinically Significant Urinalysis Results (glycosuria, ketonuria, or proteinuria) by Treatment Group. Percentages based on number of patients with at least one non-missing post-baseline urinalysis value in each treatment group. Patients are only counted once per criterion per laboratory test. The number of participants with potential clinical important urinalysis findings at any post-baseline visit were reported.
Time Frame: Immediately post-baseline up to Week 12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID | 37.5 mg BID Dexpramipexole | 75 mg BID Dexpramipexole | 150 mg BID Dexpramipexole
Number analyzed (Participants) | 27 | 22 | 26 | 28
Participants
  glycosuria (glucose in urine ++++) | 1 | 2 | 1 | 0
  ketonuria (ketones in urine ≥ ++++) | 0 | 0 | 0 | 0
  proteinuria (protein in urine ≥ ++) | 1 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Potentially Clinically Significant Vital Signs Results by Treatment Group Post Randomization Through Week 12
Description: Number of Participants with Potentially Clinically Significant Vital Signs Results by Treatment Group. Percentages based on number of patients with at least one non-missing post-baseline value in each treatment group. Patients are only counted once per criterion per laboratory test.
Time Frame: Immediately post-baseline up to Week 12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID | 37.5 mg BID Dexpramipexole | 75 mg BID Dexpramipexole | 150 mg BID Dexpramipexole
Number analyzed (Participants) | 27 | 22 | 26 | 28
Participants
  Systolic blood pressure: >180 mmHg | 0 | 0 | 0 | 0
  Systolic blood pressure: Increase >40 mmHg | 0 | 0 | 0 | 0
  Systolic blood pressure: <90 mmHg | 0 | 0 | 0 | 0
  Systolic blood pressure: Decrease >30 mmHg | 0 | 0 | 0 | 0
  Diastolic blood pressure: >105 mmHg | 0 | 0 | 0 | 0
  Diastolic blood pressure: Increase >30 mmHg | 0 | 1 | 0 | 0
  Diastolic blood pressure: <50 mmHg | 0 | 0 | 0 | 0
  Diastolic blood pressure: Decrease >20 mmHg | 0 | 0 | 0 | 0
  Pulse: >120 bpm | 0 | 0 | 0 | 0
  Pulse: Increase >30 bpm | 0 | 0 | 0 | 0
  Pulse: <50 bpm | 0 | 1 | 0 | 0
  Pulse: Decrease >20 bpm | 0 | 0 | 1 | 1
  Temperature: >38.5°C and an increase ≥1°C | 0 | 0 | 0 | 0
  Body weight: Increase ≥7% from Baseline | 0 | 0 | 1 | 1
  Body weight: Decrease ≥7% from Baseline | 0 | 0 | 0 | 1

10. Secondary Outcome: Number of Participants With Potentially Clinically Significant ECG Results by Treatment Group Post Randomization Through Week 12
Description: Number of Participants with Potentially Clinically Significant ECG Results by Treatment Group. Percentages based on number of patients with at least one non-missing post-baseline value in each treatment group. Patients are only counted once per criterion per laboratory test.
Time Frame: Immediately post-baseline up to Week 12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo BID | 37.5 mg BID Dexpramipexole | 75 mg BID Dexpramipexole | 150 mg BID Dexpramipexole
Number analyzed (Participants) | 27 | 22 | 26 | 28
Participants
  Heart Rate >120 bpm | 0 | 0 | 0 | 0
  Heart Rate Increase from Baseline >30 bpm | 0 | 0 | 0 | 1
  QT Interval: >450 ms | 0 | 0 | 0 | 0
  QT Interval: >480 ms | 0 | 0 | 0 | 0
  QT Interval: >500 ms | 0 | 0 | 0 | 0
  QT Interval: Increase from Baseline >30 ms | 7 | 3 | 2 | 0
  QT Interval: Increase from Baseline >60 ms | 0 | 0 | 0 | 0
  QTcF Interval: >450 ms | 0 | 0 | 0 | 0
  QTcF Interval: >480 ms | 0 | 0 | 0 | 0
  QTcF Interval: >500 ms | 0 | 0 | 0 | 0
  QTcF Interval: Increase from Baseline >30 ms | 1 | 0 | 0 | 0
  QTcF Interval: Increase from Baseline >60 ms | 0 | 0 | 0 | 0
  Change from Baseline in PR >25% and PR value >220 ms | 0 | 0 | 0 | 0
  Change from Baseline in QRS >25% and QRS value >110 ms | 0 | 0 | 0 | 0

11. Other Pre Specified Outcome: Change in Nasal Eosinophil Peroxidase (Presented as Ratio to Protein) From Baseline to Week 12
Description: The EPX:protein ratio was used to normalize the EPX for the quantity of sample, yielding the values in ng EPX per mg protein. The ratio of nasal Eosinophil Peroxidase to Protein is a biomarker for airway eosinophils. A lower ratio to Baseline represents a lowering in airway eosinophilia, which is a marker of successful drug therapy.
Time Frame: Baseline, Week 12
Population: The efficacy population was a modified intent-to-treat sample and consists of all subjects in the safety population (all subjects who were randomized and received at least one dose of randomized study drug) and who had both Baseline (non-zero) and Week 12 values.
Measure: Median (Inter-Quartile Range); unit: ratio to baseline
Arm/Group | Placebo BID | 37.5 mg BID Dexpramipexole | 75 mg BID Dexpramipexole | 150 mg BID Dexpramipexole
Number analyzed (Participants) | 15 | 16 | 19 | 19
ratio to baseline | 0.833 [0.258 to 2.99] | 0.645 [0.275 to 1.18] | 0.174 [0 to 0.708] | 0.110 [0 to 0.943]
Statistical Analysis 1: Comparison: Placebo BID vs 150 mg BID Dexpramipexole; The 150 mg BID dexpramipexole group was compared to placebo at Week 12 using a Wilcoxon rank sum test; Test type: Superiority; p = 0.0196, Wilcoxon (Mann-Whitney) — No adjustment for multiple testing of exploratory endpoints was used
Statistical Analysis 2: Comparison: Placebo BID vs 75 mg BID Dexpramipexole; The 75mg BID dexpramipexole group was compared to placebo at Week 12 using a Wilcoxon rank sum test; Test type: Superiority; p = 0.0207, Wilcoxon (Mann-Whitney) — No adjustment for multiple testing of exploratory endpoints was used
Statistical Analysis 3: Comparison: Placebo BID vs 37.5 mg BID Dexpramipexole; The 37.5 mg BID dexpramipexole group was compared to placebo at Week 12 using a Wilcoxon rank sum test; Test type: Superiority; p = 0.5399, Wilcoxon (Mann-Whitney) — No adjustment for multiple testing of exploratory endpoints was used

12. Other Pre Specified Outcome: Change in Blood Absolute Blood Basophil Count From Baseline to Week 12
Description: The analysis used a mixed effects model repeated-measures MMRM with terms for baseline, GINA treatment step, treatment, visit, treatment by visit interaction, and baseline by visit interaction as fixed effects, and subject as a random effect. An unstructured covariance matrix was used. The response variable was the post-baseline value minus the baseline value. Basophils were enumerated as part of the WBC automated differential performed by the Central Laboratory.
Time Frame: Baseline, Week 12
Population: The efficacy population was a modified intent-to-treat sample and consists of all subjects in the safety population (all subjects who were randomized and received at least one dose of randomized study drug) and who have at least one post-randomization evaluation.
Measure: Least Squares Mean (Standard Error); unit: cells (10*9/L)
Arm/Group | Placebo BID | 37.5 mg BID Dexpramipexole | 75 mg BID Dexpramipexole | 150 mg BID Dexpramipexole
Number analyzed (Participants) | 25 | 22 | 24 | 28
cells (10*9/L) | -0.00439 (0.006323) | -0.00655 (0.006674) | -0.0250 (0.006487) | -0.0277 (0.006082)
Statistical Analysis 1: Comparison: Placebo BID vs 150 mg BID Dexpramipexole; The 150 mg BID dexpramipexole group was compared to placebo using a mixed effects model repeated-measures (MMRM) with terms for baseline, GINA treatment step, treatment, visit, treatment by visit interaction, and baseline by visit interaction as fixed effects, and subject as a random effect. An unstructured covariance matrix was used. The response variable was the post-baseline value minus the baseline value; Test type: Superiority; p = 0.0084, Mixed Models Analysis — No adjustment for multiple testing of exploratory endpoints was used; Mean Difference (Final Values) = -0.0233, 95% CI 2-sided [-0.0405 to -0.00613] — Estimate is the difference of the 150 mg BID group from the placebo group in the change absolute basophil count (automated differential) from Baseline to Week 12 (end of primary treatment period). A negative value represents fewer basophils
Statistical Analysis 2: Comparison: Placebo BID vs 75 mg BID Dexpramipexole; The 75 mg BID dexpramipexole group was compared to placebo using a mixed effects model repeated-measures (MMRM) with terms for baseline, GINA treatment step, treatment, visit, treatment by visit interaction, and baseline by visit interaction as fixed effects, and subject as a random effect. An unstructured covariance matrix was used. The response variable was the post-baseline value minus the baseline value; Test type: Superiority; p = 0.0237, Mixed Models Analysis — No adjustment for multiple testing of exploratory endpoints was used; Mean Difference (Final Values) = -0.0206, 95% CI 2-sided [-0.0384 to -0.00281] — Estimate is the difference of the 75 mg BID group from the placebo group in the change absolute basophil count (automated differential) from Baseline to Week 12 (end of primary treatment period). A negative value represents fewer basophils
Statistical Analysis 3: Comparison: Placebo BID vs 37.5 mg BID Dexpramipexole; The 37.5 mg BID dexpramipexole group was compared to placebo using a mixed effects model repeated-measures (MMRM) with terms for baseline, GINA treatment step, treatment, visit, treatment by visit interaction, and baseline by visit interaction as fixed effects, and subject as a random effect. An unstructured covariance matrix was used. The response variable was the post-baseline value minus the baseline value; Test type: Superiority; p = 0.8140, Mixed Models Analysis — No adjustment for multiple testing of exploratory endpoints was used; Mean Difference (Final Values) = -0.00215, 95% CI 2-sided [-0.0203 to 0.0160] — Estimate is the difference of the 37.5 mg BID group from the placebo group in the change absolute basophil count (automated differential) from Baseline to Week 12 (end of primary treatment period). A negative value represents fewer basophils

13. Other Pre Specified Outcome: Change in Fractional Exhaled Nitric Oxide (FeNO) From Baseline to Week 12
Description: FeNO is non-invasive biomarker of airway inflammation in asthma participants.
Time Frame: Baseline, Week 12
Population: as for outcome 12
Measure: Least Squares Mean (Standard Error); unit: parts per billion
Arm/Group | Placebo BID | 37.5 mg BID Dexpramipexole | 75 mg BID Dexpramipexole | 150 mg BID Dexpramipexole
Number analyzed (Participants) | 17 | 17 | 20 | 23
parts per billion | 3.38 (4.6447) | -6.79 (4.7849) | -3.14 (4.3651) | -4.86 (4.2175)
Statistical Analysis 1: Comparison: Placebo BID vs 150 mg BID Dexpramipexole; [analysis description as in outcome 12, analysis 1]; Test type: Superiority; p = 0.1886, Mixed Models Analysis — No adjustment for multiple testing of exploratory endpoints was used; Mean Difference (Final Values) = -8.24, 95% CI 2-sided [-20.6 to 4.13] — Estimate is the difference of the 150 mg BID group from the placebo group in the change in FeNO from Baseline to Week 12 in liters. In eosinophilic asthma, a lower FeNO indicates less eosinophilic inflammation of the airway than a higher value
Statistical Analysis 2: Comparison: Placebo BID vs 75 mg BID Dexpramipexole; The 75mg BID dexpramipexole group was compared to placebo using a mixed effects model repeated-measures (MMRM) with terms for baseline, GINA treatment step, treatment, visit, treatment by visit interaction, and baseline by visit interaction as fixed effects, and subject as a random effect. An unstructured covariance matrix was used. The response variable was the post-baseline value minus the baseline value; Test type: Superiority; p = 0.3061, Mixed Models Analysis — No adjustment for multiple testing of exploratory endpoints was used; Mean Difference (Final Values) = -6.53, 95% CI 2-sided [-19.1 to 6.08] — Estimate is the difference of the 75 mg BID group from the placebo group in the change in FeNO from Baseline to Week 12 in liters. In eosinophilic asthma, a lower FeNO indicates less eosinophilic inflammation of the airway than a higher value
Statistical Analysis 3: Comparison: Placebo BID vs 37.5 mg BID Dexpramipexole; [analysis description as in outcome 12, analysis 3]; Test type: Superiority; p = 0.1294, Mixed Models Analysis — No adjustment for multiple testing of exploratory endpoints was used; Mean Difference (Final Values) = -10.2, 95% CI 2-sided [-23.4 to 3.04] — Estimate is the difference of the 37.5 mg BID group from the placebo group in the change in FeNO from Baseline to Week 12 in liters. In eosinophilic asthma, a lower FeNO indicates less eosinophilic inflammation of the airway than a higher value

ADVERSE EVENTS:
Time Frame: Placebo Run-in Period = from enrollment to Randomization (2-4 weeks); Primary Assessment Period = from Randomization through the Week 12 visit, plus 30 days following the last dose; Eosinophil Recovery Period = all visits occurring from 30 days following the last dose through the end of study (Week 24 post-Randomization)
Groups:
- Screening Period: All subjects who signed informed consent and entered the Primary Assessment Period
- Primary Assessment Period: Placebo BID: Following the 2-4 week placebo Run-in Period, randomized subjects continued to receive 1 tablet placebo twice daily for 12 weeks during the Primary Assessment Period.
  Placebo: 1 placebo tablet twice daily
- Primary Assessment Period: 37.5 mg BID: Following the 2-4 week placebo Run-in Period, randomized subjects received 1 tablet dexpramipexole 37.5 mg twice daily for 12 weeks during the Primary Assessment Period.
  Dexpramipexole: 1 dexpramipexole tablet twice daily
- Primary Assessment Period: 75 mg BID: Following the 2-4 week placebo Run-in Period, randomized subjects received 1 tablet dexpramipexole 75 mg twice daily for 12 weeks during the Primary Assessment Period.
  Dexpramipexole: 1 dexpramipexole tablet twice daily
- Primary Assessment Period: 150 mg BID: Following the 2-4 week placebo Run-in Period, randomized subjects received 1 tablet dexpramipexole 150 mg twice daily for 12 weeks during the Primary Assessment Period.
  Dexpramipexole: 1 dexpramipexole tablet twice daily
- Eosinophil Recovery Period: Assigned to Placebo BID During Primary Assessment Period; Eosinophil Recovery Period: Assigned to 37.5 mg BID During Primary Assessment Period; Eosinophil Recovery Period: Assigned to 75 mg BID During Primary Assessment Period; Eosinophil Recovery Period: Assigned to 150 mg BID During Primary Assessment Period: Following the Primary Assessment Period, subjects were followed within their randomized treatment group
Arm/Group | Screening Period | Primary Assessment Period: Placebo BID | Primary Assessment Period: 37.5 mg BID | Primary Assessment Period: 75 mg BID | Primary Assessment Period: 150 mg BID | Eosinophil Recovery Period: Assigned to Placebo BID During Primary Assessment Period | Eosinophil Recovery Period: Assigned to 37.5 mg BID During Primary Assessment Period | Eosinophil Recovery Period: Assigned to 75 mg BID During Primary Assessment Period | Eosinophil Recovery Period: Assigned to 150 mg BID During Primary Assessment Period
All-Cause Mortality (participants affected / at risk) | 0/103 | 0/27 | 0/22 | 0/26 | 0/28 | 0/25 | 0/22 | 0/24 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/103 | 0/27 | 0/22 | 0/26 | 0/28 | 0/25 | 0/22 | 0/24 | 0/28
Other Adverse Events (participants affected / at risk) | 6/103 | 9/27 | 7/22 | 12/26 | 12/28 | 2/25 | 3/22 | 5/24 | 10/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Screening Period (N=103) | Primary Assessment Period: Placebo BID (N=27) | Primary Assessment Period: 37.5 mg BID (N=22) | Primary Assessment Period: 75 mg BID (N=26) | Primary Assessment Period: 150 mg BID (N=28) | Eosinophil Recovery Period: Assigned to Placebo BID During Primary Assessment Period (N=25) | Eosinophil Recovery Period: Assigned to 37.5 mg BID During Primary Assessment Period (N=22) | Eosinophil Recovery Period: Assigned to 75 mg BID During Primary Assessment Period (N=24) | Eosinophil Recovery Period: Assigned to 150 mg BID During Primary Assessment Period (N=28)
Monocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Sinus Bradycardia (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Corona virus infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear infection fungal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1 | 3 | 0 | 1 | 1 | 0 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Urethritis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Foreign body in ear (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Coronavirus test positive (Investigations) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
Fluid retention (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0 | 2 | 1 | 1 | 0 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Eye contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Knopp's agreements with its investigators may vary. However, Knopp does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial, and are subject to a minimum 60 day review period by Knopp.

DOCUMENTS (2):
  • Study Protocol (2019-07-16): https://cdn.clinicaltrials.gov/large-docs/39/NCT04046939/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/39/NCT04046939/SAP_001.pdf